CLINICAL TRIAL: NCT06661057
Title: Avation Electric Stimulation System for Spinal Cord Injury Neurogenic Bladder: A Hybrid Effectiveness-implementation Pilot Trial
Brief Title: Avation Electric Stimulation System for Spinal Cord Injury Neurogenic Bladder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Industry partner decided not proceed
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Mission Connect (Unknown)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-0834
Record Dates: First submitted 2024-10-15; First posted 2024-10-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Neurogenic Bladder
Keywords: spinal cord injury; tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vivally system (Experimental)
  Interventions: Device: Vivally system stimulation

INTERVENTIONS:
Device: Vivally system stimulation — During the first month, participants will do the stimulation at different time points: 1) supine while in bed, 2) seated in the morning, 3) sitting in the afternoon, and 4) sitting in the evening. Participants will measure the circumference of their ankle prior to each use. Participants will use the System for an additional 2 months with the preferred stimulation parameters based on the study team's recommendations from the first month of use.

SUMMARY:
The purpose of this study is to assess and optimize the Avation electric stimulation system output and electromyography (EMG) processing to stimulate the tibial nerve in people with chronic Spinal Cord Injury (SCI) who have foot muscle atrophy and edema, both of which may affect proper device operations, to evaluate the safety, feasibility, and effectiveness of Avation Electric Stimulation System for bladder neuromodulation in people with SCI and identify barriers to implementation of the existing Avation Electric Stimulation System to help with developing it towards a new indication for routine care of SCI NB.

ELIGIBILITY:
Inclusion Criteria:

* Injury level above T10.
* Diagnosis of neurogenic bladder (Performing intermittent catheterization).
* English or Spanish Speaker.
* Toe flexion upon tibial nerve stimulation with transcutaneous electric stimulation.
* No adverse events during the Vivally 5-minute trial

Exclusion Criteria:

* Intradetrusor Botulinum Toxin within six months.
* Presence of urinary tract infection (UTI) symptoms.
* Pregnancy or breastfeeding.
* Known allergy to electrode or device materials.
* Known intolerance to leg electric stimulation
* Patient with no smartphone access.
* Pain/discomfort or adverse reaction with the trial of toe flexion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Consistency and Reliability of Stimulation Output as assessed by the percentage of sessions where the desired stimulation intensity is achieved (based on EMG waveform consistency) and time of day (morning, afternoon, evening) | Daily during the 4-week optimization period
EMG Waveform Quality as assessed by the number of successful EMG detections per session versus unsuccessful ones | Daily during the 4-week optimization period
Safety as assessed by the Pain score reported on the participant diary | Continuous, daily monitoring throughout the 12-week study
  Pain is scored on linear scale from 0(no pain)-10(worst pain), higher score indicating worse outcome
Safety as assessed by the adverse events self reported by participant | Continuous, daily monitoring throughout the 12-week study
  patient-reported adverse events, including changes in spasticity, their bowel programs, urinary tract infections, autonomic dysreflexia, and all other concerning changes
Feasibility as assessed by the number of participants who adhere to the protocol as reported on the patient dairy | Weekly during the 12-week study
Effectiveness for Bladder Control as assessed by the changes in volume of catheterization reported in the voiding diary data | 2 days per month for all three months
Effectiveness for Bladder Control as assessed by the changes in frequency of catheterization reported in the voiding diary data | 2 days per month for all three months
Effectiveness for Bladder Control as assessed by the number of episodes of incontinence reported in the voiding diary data | 2 days per month for all three months
Effectiveness for Bladder Control as assessed by the changes in volume of catheterization reported in the voiding diary data | Once a month for all 3 months
Effectiveness for Bladder Control as assessed by the changes in frequency of catheterization reported in the voiding diary data | Once a month for all 3 months
Effectiveness for Bladder Control as assessed by the number of episodes of incontinence reported in the voiding diary data | Once a month for all 3 months
Implementation Barriers as assessed by a survey | end of study (12 weeks from baseline)
Patient-Reported Implementation Feedback as assessed by a survey | end of study (12 weeks from baseline)

SECONDARY OUTCOMES:
Patient-Reported Comfort as assessed by the participant survey | Daily during the 4-week optimization period
Patient-Reported Usability as assessed by the participant survey | Daily during the 4-week optimization period
Type and extent of adjustments (none, minor, major) required for System Operation needed for effective stimulation | End of the 4-week optimization period
Frequency of adaptations made to the device | End of the 4-week optimization period
Number of participants that had adaptations made to the device as assessed by a yes or no questionnaire | End of the 4-week optimization period
Change in Quality of Life as assessed by the The Neurogenic Bladder Symptom Score (NBSS) | Baseline, 4 weeks, 8 weeks and 12 weeks
  This is a 24 item questionnaire that measures bladder symptoms across 3 different domains: incontinence (scored 0-29), storage and voiding (scored 0-22), and consequences (scored 0-23) for a maximum score of 74, higher scores indicating worse outcome
Change in Quality of Life as assessed by the Incontinence Quality of Life Questionnaire(I-QOL) | Baseline, 4 weeks, 8 weeks and 12 weeks
  The I-QOL is a 22-item self-reported questionnaire scored on a scale from 0 to 100, with higher scores indicating better quality of life.
Change in Quality of Life as assessed by the Neurogenic Bowel Dysfunction (NBD) score | Baseline, 4 weeks, 8 weeks and 12 weeks
  The NBD score evaluates symptoms such as incontinence, constipation, and frequency of bowel management interventions. It is scored on a scale from 0 to 47, with higher scores indicating more severe dysfunction.
Patient satisfaction as assessed by a survey | End of study (12 weeks form baseline)
  This is an 8 item questionnaire and each is scored between 1(strongly disagree)-5( strongly agree),maximum score of 40, higher score indicates better satisfaction with the device
Qualitative assessment of edema or skin changes as assessed by photos of lower leg and foot | Weekly during the 12-week study
Patient-Reported Changes in Bladder Program | Weekly during the 12-week study
  Documentation of any changes made to the bladder management program
Number of caregivers who were satisfied as assessed by the interview | end of study (12 weeks from baseline)
Number of clinicians who were satisfied as assessed by the interview | end of study (12 weeks from baseline)
System Fidelity as assessed by the degree to which the the Avation electric stimulation system was used as intended by patients | end of study (12 weeks from baseline)
  This is assessed by the the number of times participant used the device per month
Relative Advantage and Adaptability of the Innovation as assessed by the ratings on the perceived benefits and adaptability of the the Avation electric stimulation system compared to existing treatments | end of study (12 weeks from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, MS, Principal Investigator — The University of Texas Health Science Center and Houston

IPD SHARING:
Plan to Share IPD: No